CLINICAL TRIAL: NCT04583241
Title: Prospective Study of Patients Treated for Bone and Joint Infection (BJI) Due to Staphylococcus Aureus, Aiming at Identifying Biomarkers of Diagnosis Interest in Chronic BJI
Acronym: ESPRI-IOAC
Status: Terminated | Type: Observational
Why Stopped: difficulties in including patients with Staphylococcus aureus infection
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL20_0235
Record Dates: First submitted 2020-10-05; First posted 2020-10-12 (Actual); Last update posted 2022-06-23 (Actual); Status verified 2022-06

CONDITIONS: Bone and Join Infection (BJI); Periprosthetic Joint Infection (PJI)
Keywords: BJI; Staphylococcus aureus; biomarkers
MeSH Terms: conditions — Staphylococcal Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * Collection of serum : Blood samples are obtained at different times : Day 0 (day of surgery), and for patients with staphylococcus aureus monoinfection who are follow-up during two years, at week 2, week 6 post-surgery, at the end of antibiotherapy and 6 months post-surgery)
  * Tissue bank : Recovery of residual samples of bone tissue, joint fluid, fragment of prostheses the day of surgery
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- BJI group: Patients with an BJI on material (prosthesis or other implant) infected by Staphylococcus aureus* Patients are follow-up during two years after surgery.
  *Diagnosis of staphylococcus aureus monoinfection realized a posteriori after surgery on bacteriological sample
  Interventions: Other: Constitution of serum bank at D0; Other: Constitution of serum bank during follow-up; Other: ELISA assays of serum markers of bone remodeling at D0; Other: ELISA assays of serum markers of bone remodeling during follow-up; Other: Analysis of bacterial gene expression at D0
- Control Group With material: Patients with mechanical problems on implanted equipment (control cohort), without infection* Patient of this group are follow-up until surgery.
  *Diagnosis of staphylococcus aureus monoinfection realized a posteriori after surgery on bacteriological sample
  Interventions: Other: Constitution of serum bank at D0; Other: ELISA assays of serum markers of bone remodeling at D0; Other: Analysis of bacterial gene expression at D0
- Group osteomyelitis: Patients with chronic osteomyelitis* Patient of this group are follow-up until surgery.
  *Diagnosis of staphylococcus aureus monoinfection realized a posteriori after surgery on bacteriological sample
  Interventions: Other: Constitution of serum bank at D0; Other: ELISA assays of serum markers of bone remodeling at D0; Other: Analysis of bacterial gene expression at D0
- Control Group with cruciate ligament surgery: Patients having cruciate ligament surgery Patient of this group are follow-up until surgery.
  Interventions: Other: Constitution of serum bank at D0; Other: ELISA assays of serum markers of bone remodeling at D0; Other: Analysis of bacterial gene expression at D0

INTERVENTIONS:
Other: Constitution of serum bank at D0 — Blood samples at Day 0 (day of surgery)
Other: Constitution of serum bank during follow-up — Blood samples are obtained at week 2, week 6 post-surgery, at the end of antibiotherapy and 6 months post-surgery, only for patients with staphylococcus aureus monoinfection who are follow-up during two years.
  Groups: BJI group
Other: ELISA assays of serum markers of bone remodeling at D0 — Assessment by ELISA assays of serum markers of bone remodelling: the osteocalcin (OC), the procollagen propeptide type 1 (PINP), the cross linked telopeptide of type 1 collagen (CTX1) and the periostin at Day 0 (day of surgery)
Other: ELISA assays of serum markers of bone remodeling during follow-up — Assessment by ELISA assays of serum markers of bone remodelling: the osteocalcin (OC), the procollagen propeptide type 1 (PINP), the cross linked telopeptide of type 1 collagen (CTX1) and the periostin at week 2, week 6 post-surgery, at the end of antibiotherapy and 6 months post-surgery, only for patients with staphylococcus aureus monoinfection who are follow-up during two years
  Groups: BJI group
Other: Analysis of bacterial gene expression at D0 — Assessement of bacterial gene expression on surgery residual tissue (bone tissue, joint fluid, fragment of prostheses) collected at Day 0 (day of the surgery)

SUMMARY:
There are more than one million (> 40,000 cases per year in France) of osteoarticular infections (OAI) yearly in the world. The number of these infections is constantly increasing due to an increase in life expectancy associated with an increase in prosthesis fitting, as well as an increase in comorbid factors. These are severe pathologies associated with mortality (5%) and significant morbidity (40%), responsible for functional sequelae with an individual cost (prolonged hospitalization, altered quality of life, disability) and societal (sick leave, partial disability). or total, temporary or permanent) extremely high. In addition, reinfection rates within two years of treatment are high.

The BJIs are a group of clinical entities that have in common the invasion and progressive destruction of bone and cartilage tissue by bacterial-like microorganisms.

Staphylococcus spp is the main pathogen (>50%) in BJI and is associated with particularly difficult to treat infections, with a high rate of chronicity and relapses, especially in case of implanted material.

The difficulty in managing these infections is partly linked, on the one hand, to the fact that the pathogens are in "persistent" metabolic forms and in intracellular reservoirs which make them insensitive to conventional antibiotics and, on the other hand, the absence of reliable markers of the infection and above all of its clinical resolution, which complicates clinical trials.

ESPRI-IOAC is a consortium of 4 partners (private-public) from Lyon area and which aims at:

* studying the translational value of BJI preclinical models
* identifying biomarkers of infection in preclinical models and at assessing them in a prospective study.

The current study is part of the global ESPRI-IOAC consortium, and represent the clinical application.

It is a prospective study of patients treated for BJI in the infectious disease department of the Hospices Civils de Lyon, La Croix-Rousse, for osteo-articular infections due to Staphylococcus aureus, or for simple mechanical revision or for cruciate ligament surgery, the objective of which is to highlight biomarkers of interest in the diagnosis of chronic BJI and, or predictive of the therapeutic response.

The translational value of the experimental models used in the BJI will also be studied.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 30 years old
* Hospitalized in orthopedic surgery for one of these reasons:
* A suspected infection or a documented proven infection with staphylococcus aureus on prosthesis or other orthopedic implant
* A mechanical cause (absence of infection) on prosthesis or orthopedic implant
* Documented chronic osteomyelitis due to staphylococcus aureus
* Cruciate ligament surgery
* Patient not subject to any legal protection measure
* Patient who can be followed in the Infectious and Tropical Diseases Department, CRIOAC Lyon ("Centre de Référence des Infections Ostéo-Articulaires complexes" = reference centre of bone and joint infections in french), La Croix-Rousse for at least 6 months post-surgery
* Patient who gave his no-opposition
* Patient giving his consent to the creation of biological collections

Exclusion Criteria:

* Polymicrobial infection
* Known inflammatory disease
* Hyperthyroidism
* Cushing's disease
* Osteomalacia
* Renal osteodystrophy
* Paget's disease
* Malignant disease in progress
* Multiple myeloma
* Bone metastases
* Ehlers-Danlos syndrome
* Pregnant or lactating woman
* Renal impairment (Creatinine clearance <60 mL / min)
* Trauma in the 6 months preceding surgery
* Fracture in the 6 months preceding surgery
* Corticosteroid therapy in progress at the time of inclusion
* Active infection with HIV (human immunodeficiency virus), HBV (hepatitis B virus), HCV hepatitis C virus) documented in the patient file
* Antibiotic treatment in the 15 days preceding inclusion
* People placed under judicial protection

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated in the orthopedic surgery and infectious diseases departments of the Hospices Civils de Lyon, Croix-Rousse Hospital, for osteo-articular infections, due to Staphylococcus aureus, for simple mechanical revision or for cruciate ligament surgery.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2020-11-27 (Actual); Primary Completion 2022-01-26 (Actual); Study Completion 2022-01-26 (Actual)

PRIMARY OUTCOMES:
Dosages of serum osteocalcin | At the time of surgery
  Comparison of dosages by ELISA test of serum osteocalcin between the patients with OAI and the "control" patients without OAI at the time of inclusion in order to demonstrate a marker or a combination of markers for OAI.
Dosages of serum procollagen propeptide type 1 | At the time of surgery
  Comparison of dosages by ELISA test of serum procollagen propeptide type 1 between the patients with OAI and the "control" patients without OAI at the time of inclusion in order to demonstrate a marker or a combination of markers for OAI.
Dosages of serum cross-linked telopeptide of type 1 collagen | At the time of surgery
  Comparison of dosages by ELISA test of serum cross-linked telopeptide of type 1 collagen between the patients with OAI and the "control" patients without OAI at the time of inclusion in order to demonstrate a marker or a combination of markers for OAI.
Dosages of serum periostin | At the time of surgery
  Comparison of dosages by ELISA test of serum periostin between the patients with OAI and the "control" patients without OAI at the time of inclusion in order to demonstrate a marker or a combination of markers for OAI.

CONTACTS AND LOCATIONS:
Overall Officials: Tristan FERRY, Pr, Principal Investigator — Service Maladies Infectieuses et Tropicales, CRIOAC Lyon
Locations (1):
- Hôpital Croix Rousse, Lyon, France